CLINICAL TRIAL: NCT06178276
Title: Investigation of Neurophysiological Functioning During Oral Comprehension Task. An Exploratory Study in Second Language (Italian) Learning in French Students Using Autonomic and Cerebral Investigation
Brief Title: Investigation of Neurophysiological Functioning During Oral Comprehension Task
Acronym: COraIL
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Grenoble Alps (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 38RC23.0309; 2023-A01939-36 (Other: ID RCB)
Record Dates: First submitted 2023-11-16; First posted 2023-12-20 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Learning; Language; Comprehension
Keywords: Language Learning; Oral comprehension; autonomic activity; brain activity
MeSH Terms: conditions — Language | interventions — Microbial Interactions; Diagnostic Imaging; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A2 level: Level of oral comprehension in italian language
  Interventions: Diagnostic Test: behavior; Diagnostic Test: physiology; Diagnostic Test: imaging
- B2 level: Level of oral comprehension in italian language
  Interventions: Diagnostic Test: behavior; Diagnostic Test: physiology; Diagnostic Test: imaging

INTERVENTIONS:
Diagnostic Test: behavior — behavioral measurements will be performed during the oral comprehension testing
Diagnostic Test: physiology — physiologic (autonomic) measurements will be performed during the oral comprehension testing
  Other Names: autonomic
Diagnostic Test: imaging — central (brain) measurements will be performed during the oral comprehension testing
  Other Names: fMRI

SUMMARY:
The oral comprehension (OC) of a second language (L2) involves different cognitive processes, specially during the learning phase. This study aims at investigating the neurophysiological functioning of different steps involved in this oral understanding.

DETAILED DESCRIPTION:
Here, the investigators seek for the different neurophysiological processes involved in OC according to the level of understanding (2 levels) and its different phases (fluid, hindered and metacognitive feedback).

This study therefore requires three different research methodologies :

1. an interactive system dedicated to the boundary delimitations of obstacles during OC
2. an investigation of the autonomic nervous system responses (measurement of electrodermal activity and heart rate variability) that will likely occur differently during different phases of the OC process
3. an investigation of the central responses (through fMRI technique), coupled with autonomous responses, that will identify the different neural networks in the different stages of the OC process.

ELIGIBILITY:
Inclusion Criteria:

* French learner in Italian language
* right-handed
* affiliated to French social security
* informed consent signed

Exclusion Criteria:

* pregnant woman
* audiologic pathology impacting the capacity of hearing
* neurologic or psychiatric pathology that may interfere with oral comprehension
* learning disability (for instance: dyslexia)
* contra-indication to MRI and to EDA acquisition

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: French learner in Italian language recruited at university
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Sympathetic activity | up to 3 months following the language profile completion
  ElectroDermal Activity (EDA) measured in µS

SECONDARY OUTCOMES:
Parasympathetic activity | up to 3 months following the language profile completion
  Heart Rate Variability (HRV) measured using the relative power of the high-frequency (HF) component of the HRV (in % of the total power)
Activated brain regions demonstrating brain activity | up to 6 months following the language profile completion
  fMRI brain imaging data will be analyzed using Statistical Parametric Mapping (SPM12).
Correlations between sympathetic and parasympathetic activity | up to 3 months following the language profile completion
  correlation between EDA components measured in µS and relative power of the HF-HRV
Interaction between sympathetic activity and brain activity | up to 6 months following the acquisition of language profile
  Correlation of EDA (µS) with fMRI brain imaging data
Interaction between parasympathetic activity and brain activity | up to 6 months following the acquisition of language profile
  Correlation of relative HF component of HRV with the fMRI brain imaging data
Linguistic evaluation | up to 1 month following the acquisition of language profile
  Linguistic processes are assessed by performance score on the following tests:
  verbal fluency test in first language (number of items found in 1 min)
  verbal fluency test in second language (number of items found in 1 min)
Cognitive evaluation of executive functions | up to 1 month following the acquisition of language profile
  Cognitive evaluation assessed by the following tests:
  Trail Making Test (TMT-A and TMT-B) scores. Time duration (in seconds) for each subtest. Shortest duration meaning efficient executive functions
Cognitive evaluation of short term memory | up to 1 month following the acquisition of language profile
  WAIS4 subtest (measured by scores)

CONTACTS AND LOCATIONS:
Overall Officials: Triscia Biagiotti, Ms, Study Chair — University Grenoble Alpes
Locations (1):
- University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided
anonymised, processed data will be shared after publication acceptance on dedicated sites